CLINICAL TRIAL: NCT04700657
Title: Investigation of the Prevalence of Hypoesthesia Related Neurotrophic Keratitis in Patients With Ocular Graft Versus Host Disease
Brief Title: The Prevalence of Hypoesthesia Related Keratitis in Ocular Graft Vs. Host Disease (GVHD) Patients
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shaohui Liu, Principal Investigator, Indiana University
Other Study IDs: 2004207079
Record Dates: First submitted 2020-11-23; First posted 2021-01-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Ocular GVHD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 15 patients affected by ocular GVHD
  Interventions: Diagnostic Test: corneal sensation test
- 15 age-matched normal volunteers.
  Interventions: Diagnostic Test: corneal sensation test

INTERVENTIONS:
Diagnostic Test: corneal sensation test — Thorough ocular surface study including corneal sensation test in the GVHD group, comparing to the normal control group

SUMMARY:
The Investigators hypothesize that the recalcitrant nature of ocular GVHD may be related to corneal nerve damage and corneal hypoesthesia. The investigators aim to study the prevalence of corneal hypoesthesia in GVHD patients and its correlation with ocular surface changes.

DETAILED DESCRIPTION:
Rationale: Graft-versus-host disease(GVHD) is a common complication of allogeneic bone marrow or hematopoietic stem cell transplantation (HSCT). It affects multiple systems, including skin, gastrointestinal system, liver, lung, and oral cavity, as well as eyes, which contributes to decreased quality of life and increased mortality. About 10% of patients with acute GVHD and 60-90% of those with chronic GVHD develop ocular complications. Dry eye is the most common manifestation of ocular GVHD. The pathogenesis remains unclear. The conjunctival tissue and cornea are the main immunological targets in GVHD. Patients often have punctate hypothesize that the recalcitrant nature of ocular GVHD may be related to corneal nerve damage and sensation changes.

There are a few confocal microscopy studies on corneal nerve changes in GVHD, including increased tortuosity and reduced reflectivity of sub-basal nerves. However, there were very few studies on clinical correlations of those microscopic changes with corneal sensation and ocular surface health. In addition, confocal microscopes are not widely available in clinical practice. It also requires the special expertise of technicians and physicians to obtain and explain the images. It is therefore not feasible to routinely perform confocal microscopy for corneal innervation study.

The investigators plan to study the corneal sensation changes and their correlation with ocular surface staining, tear film breakdown and meibomian gland dysfunction in GVHD patients. The study will shed light on an important aspect of corneal innervation damage in GVHD and may lead to new treatment modalities for those patients, noting that topical recombinant human nerve growth factor cenegermin was recently FDA approved for neurotrophic keratopathy. The investigators intend to identify the ocular characteristics of GVHD patients that may potentially benefit from cenegermin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic GVHD is diagnosed based on the history of allogeneic HSCT (Hematopoietic stem cell transplant) and the presence of systemic GVHD in organs other than the eye. In the ocular GVHD group, dry eye symptoms start after the development of systemic GVHD. If post-HSCT dry eye precedes GVHD clinical signs in other organs, the investigators will use the 2013 diagnostic criteria by International chronic ocular GVHD consensus group.
* The investigators will recruit patients for the study. The investigators plan to include ocular GVHD patients that are of age 18 years or older who have typical symptoms of dry eye with an Ocular Surface Disease Index (OSDI) score greater than 13 and corneal fluorescein staining (CFS) score of 3 or more (National Eye Institute [NEI] grading scale, 0-15). Normal age-matched volunteer group will include people whose OSDI less or equal to 13 and CFS score less than 3.

The patients will continue their current systemic and ocular medications, which may include one or combination of preservative free artificial tears, restasis or xiidra, serum tears, ointment, or scleral contact lens.

Exclusion Criteria:

* patients with a history of herpetic simplex or zoster keratitis, ocular or neurologic surgery (including laser or refractive surgical procedure) within 3 months before enrollment, trauma, diabetes with signs of peripheral neuropathy.
* patients with active corneal thinning or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 eyes from 15 patients affected by ocular GVHD, and 30 healthy control eyes from 15 age-matched normal volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Corneal Hypoesthesia | Baseline clinic visit
  Corneal Sensation in GVHD compared to healthy age matched controls as measured with Cochet Bonet esthesiometer.

SECONDARY OUTCOMES:
dry eye questionnaire, dry eye signs, meibomian gland dysfunction | Baseline clinic visit
  1. correlation between corneal hypoesthesia and OSDI questionaire (scale 0-100 points, where higher is worse symptoms)
  2. correlation between corneal hypoesthesia and measure of tear break up time (seconds, where less is worse)
  3. correlation between corneal hypoesthesia and bulbar redness (scale 0-4 where higher is worse)
  4. correlation between corneal hypoesthesia and tear meniscus height (measured in mm where less than 0.2mm is worse)
  5. correlation between corneal hypoesthesia and meibomiography using oculus keratograph ( lower is better)
  6. correlation between corneal hypoesthesia and fluorescein staining at slit lamp (NEI scale 0-15 where higher is worse)
  7. correlation between corneal hypoesthesia and lissamine green staining (NEI scale 0-8 where higher is worse)
  8. correlation between corneal hypoesthesia and schirmer test without anesthesia (measured in mm at 5 minutes where fewer mm of wetting is worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Glick Eye Institute - Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No